CLINICAL TRIAL: NCT03941197
Title: Ready and Healthy for Kindergarten- A Family Literacy Program for Latino Families
Brief Title: A Family Literacy Program for Latino Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Manuel E. Jimenez, MD, MS, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro2019000570
Record Dates: First submitted 2019-04-18; First posted 2019-05-07 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Literacy
Keywords: child development; family literacy program; primary care
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ready and Healthy for Kindergarten Family Literacy Program (Experimental): Ready and Healthy for Kindergarten Family Literacy Program- 8 weekly parent child workshops with text message reminders
  Interventions: Behavioral: Ready and Healthy for Kindergarten Family Literacy program

INTERVENTIONS:
Behavioral: Ready and Healthy for Kindergarten Family Literacy program — Participants will participate in 8 parent-child health-themed literacy workshops. Participants will receive 2-3 text messages per week for 8 weeks.

SUMMARY:
A pilot study of a health-focused family literacy program. The program will consist of a series of 8 weekly workshops centered around different health topics (e.g. physical activity) that introduce basic literacy skills. The workshops are designed for children entering kindergarten and their parents

DETAILED DESCRIPTION:
This is a pilot study of a health-focused family literacy program. The program consists of 8 weekly health-themed workshops designed to introduce basic literacy skills to children entering Kindergarten and their parents. There will be a pre and post test assessment for participating parents and children. During the 8 weeks, parents will receive 2-3 weekly text messages to reinforce material presented at the weekly workshop.

ELIGIBILITY:
Inclusion Criteria:

* Preferred language is either Spanish or English.
* Parent or legal guardian of child
* Parent age 18 or older
* Willing to accept text messages

Exclusion Criteria:

* Children not entering Kindergarten in Fall 2019 and their parents will be excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2019-09-28 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) Questionnaire | After 8 week period.
  Acceptability will be measured using the Acceptability of Intervention Measure (AIM). The AIM consists of 4 questions that assess acceptability. Responses range from 1 (completely disagree) to 5 (completely agree). Scales are created by averaging responses.

SECONDARY OUTCOMES:
StimQ-Preschool survey | At enrollment and after 8 week period.
  Parent reported measure of the cognitive home environment for children 5 months to 6 years to assess aspects of the home environment that affect child development.
Alphabet knowledge assessment survey | At enrollment and after 8 week period.
  Alphabet knowledge will be assessed.
Sight word knowledge assessment survey | At enrollment and after 8 week period.
  Sight word knowledge will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Manuel E Jimenez, MD, MS, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Manuel E Jimenez, New Brunswick, New Jersey, United States